CLINICAL TRIAL: NCT03467568
Title: Do Humans Over-consume Salt to Improve Mood
Brief Title: Does Salt Intake Improve Mood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, David Benton, Professor, Swansea University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DB-0123-SALT
Record Dates: First submitted 2018-02-16; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Mood; Salt Intake
Keywords: Mood Salt
MeSH Terms: interventions — Sodium Chloride; Water

STUDY DESIGN:
Intervention Model Description: The study has four arms. Salt alone; salt plus water; placebo alone, placebo plus water
Who Masked: Participant, Investigator
Masking Description: Salt / placebo will be consumed by capsule under a double blind procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sodium chloride / Water (Active Comparator): The sodium chloride / water arm involves 300mg sodium chloride being consumed in a capsule and on two occasions 150ml of water being drunk
  Interventions: Dietary Supplement: Sodium Chloride; Dietary Supplement: Water
- Sodium chloride / no water (Active Comparator): A capsule containing 300mg of sodium chloride will be consumed but no water will be drunk over the morning
  Interventions: Dietary Supplement: Sodium Chloride; Biological: No water consumed
- Placebo / water (Active Comparator): A capsule containing a placebo will be consumed and on two occasions 150ml of water will be drunk
  Interventions: Other: Placebo capsule; Dietary Supplement: Water
- Placebo / no water (Placebo Comparator): A capsule containing a placebo will be consumed but no water will be drunk over the morning
  Interventions: Other: Placebo capsule; Biological: No water consumed

INTERVENTIONS:
Dietary Supplement: Sodium Chloride — 300mg sodium chloride will be provided in a capsule
  Arms: Sodium chloride / Water; Sodium chloride / no water
Other: Placebo capsule — A capsule of identical appearance to that providing salt, but not containing electrolytes, will be consumed
  Arms: Placebo / no water; Placebo / water
Dietary Supplement: Water — Twice during the morning a drink of 150ml of water will be consumed
  Arms: Placebo / water; Sodium chloride / Water
Biological: No water consumed — No water will be consumed during the monring
  Arms: Placebo / no water; Sodium chloride / no water

SUMMARY:
Humans display a preference for salt although the reasons remain unclear. The aim was to examine the hypothesis that salt may enhance mood. The study compares the drinking of water with and without electrolytes (either dissolved in water or by capsule). Mood was rated over a period of 155 minutes

DETAILED DESCRIPTION:
Study 1. 120 young adults will be were recruited. They will arrive in the laboratory at 0900 having consumed their normal breakfast. Over the morning they will reported their mood by responding to one hundred millimetre visual analogue scales anchored with the words: Composed/Anxious; Hostile/Agreeable; Elated/Depressed; Unsure/Confident; Energetic/Tired; Confused/Clearheaded. These dimensions of mood came from the factor analysis that formed the basis of the Profile of Mood State questionnaire. An overall measure of mood will be calculated. .

Randomly they will receive either a 150ml glass of water, or an equivalent volume of water containing electrolytes (in total 150mg sodium chloride and 45mg potassium chloride (Gatorade G2 Low calorie (34 kcal) Thirst Quencher, Pepsico). This drink will be consumed for a first time after 50 minutes, and a second time after 140 minutes. A estimate of habitual salt preference will be gained by responding to questions concerning the adding of salt to meals and a preference for salty foods.

Study 2: One hundred and twenty young adults will be recruited. A second study attempts to replicate the first in a double-blind trial where the taste of salt was hidden by using a capsule. . Participants will be assigned to one of four experimental conditions; 1) swallowed placebo capsules; 2) swallowed capsules containing electrolyte (300mg sodium chloride); 3) received placebo capsules and plain water; 4) received capsules containing electrolyte and plain water. Each drink will be 150ml of water. The allocation of the type of capsule will be carried out double-blind, determined by computer generated random numbers.

Otherwise the procedure will be identical to study one.

ELIGIBILITY:
Inclusion Criteria: Self declared in good health -

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Mood ratings using visual analogue scales | Up to three hours
  On a hundred millimetre scale ratings will be made of with the two ends anchored with the words Agreeable/Hostile, Confused/clearheaded; composed/anxious; depressed/elated; confident/unsure; tired/energetic. Each scales produces a score between 0 and 100. When added to create a total mood score the ratings vary between zero and six hundred with a higher score indicating a better mood

SECONDARY OUTCOMES:
Ratings of thirst | Up to three hours
  Rating made using a visual analogue scale responding to the question how thirsty do you feel right now? With a high score indicated greater thrist
Body weight | Up to three hours
  Changes in body weight over morning. Scales measuring to the nearest 10g will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Psychology, Swansea University, Swansea, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No